CLINICAL TRIAL: NCT00940277
Title: Couple-Focused Group Intervention for Women With Early-Stage Breast Cancer
Brief Title: Couple-Focused Intervention for Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Christiana Care Health Services (Other); Abington Memorial Hospital (Other); Albert Einstein College of Medicine (Other); The Cooper Health System (Other); Virtua Health (Other); City University of New York, School of Public Health (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CA-65727; R01CA078084-07 (NIH); IRB#07-831 (Other: Fox Chase Cancer Center)
Record Dates: First submitted 2009-07-14; First posted 2009-07-15 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-02

CONDITIONS: Breast Cancer
Keywords: women couples counseling groups support intervention marriage
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enhanced Couples Group (Experimental): Enhanced Couples Group: consists of eight 90-minute sessions, conducted weekly. ECG has a didactic educational content presented by the group leader or practice of specific relationship communication, relationship support, and couple-focused stress management. ECG participants are also given instruction about what types of behaviors are unsupportive and training in how to not behave in an unsupportive manner.
  Interventions: Behavioral: Group Counseling
- Support Group (Experimental): Support Group: 8 weekly 90-minute group counseling sessions. Using a standard approach to supportive therapy, the group interventionists will focus on encouraging participants to share their experiences with cancer, express their emotions related to the experience, voice problems they have in coping with the cancer, and offer support and advice to other members of the group. The co-facilitators will facilitate expression of affect and the sharing of the group's common issues related to cancer. Each session has a broad topic for discussion. Topics include communication with health care providers, issues related to occupational life, and coping with medical procedures and treatment. No formal or didactic information will be provided.
  Interventions: Behavioral: Group Counseling

INTERVENTIONS:
Behavioral: Group Counseling — Group counseling

SUMMARY:
The goal of the proposed study is to evaluate the efficacy of 2 couple-focused interventions developed to reduce the psychological distress on women and their partners during and after the breast cancer experience. The first group, an Enhanced Couple-Focused Group (ECG), incorporates cognitive-behavioral interventions (e.g., relaxation, stress management skills) as well as basic relationship communication and support skills (e.g., expressing support needs constructively). The second group, a Couples' Support Group (SG), is a non-structured group where general topics are discussed. The investigators will evaluate the impact of each group condition on patients' psychological adaptation, social and role functioning, and cancer treatment adherence. The investigators will also evaluate whether patient and partner perceptions of relationship support, relationship intimacy, stress management skills, and intervention group support mediate the groups' effects on each other's psychological adaptation.

The investigators hypothesize that ECG will have stronger positive effects on patient general and cancer-related distress and well-being than SG.

The investigators hypothesize that group support will mediate greater improvements in patient psychological functioning in both groups but that the effects of group support will be significantly stronger in SG than ECG.

ELIGIBILITY:
Inclusion Criteria:

* patient has a primary diagnosis of Stage 0 (Ductal Carcinoma in situ), 1, 2, or 3a breast cancer
* patient has had breast cancer surgery within the last twelve months
* patient and partner married or cohabitating
* patient and partner 18 years of age or older
* patient and partner speak and read English
* patient and partner can provide meaningful informed consent
* patient and partner do not have any chronic physical or cognitive illness that would preclude participation in the group sessions
* couple lives within 2 hour commuting distance to the center from which they are recruited

Exclusion criteria:

- patient is male

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 611 (Actual)
Dates: Start 2007-12; Primary Completion 2014-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Mental Health Inventory | time of consent/baseline, 1 week post-intervention, 6 months post-intervention, 12 months post-intervention
Impact of Events Scale-Revised | baseline, 1 week post-intervention, 6 mos post-intervention, 12 mos post-intervention
Well-being Subscale of the Mental Health Inventory (MHI) | baseline, 1 wk post-intervention, 6 mos post-intervention, 12 mos post-intervention

SECONDARY OUTCOMES:
Mental Outcomes Survey (MOS SF-36) | baseline, 1 wk post-intervention, 6 mos post-intervention, 12 mos post-intervention
Adherence to Chemotherapy | 1 yr follow-up
Adherence to Radiation Therapy | 1 yr follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Sharon L Manne, PhD, Principal Investigator — Fox Chase Cancer Center
Locations (5):
- United States (5):
  - Christiana Care Health System, Newark, Delaware
  - Cooper Health System, Voorhees Township, New Jersey
  - Virtua Health System, Voorhees Township, New Jersey
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania

REFERENCES:
- [Result] Manne S, Kashy DA, Siegel S, Myers Virtue S, Heckman C, Ryan D. Unsupportive partner behaviors, social-cognitive processing, and psychological outcomes in couples coping with early stage breast cancer. J Fam Psychol. 2014 Apr;28(2):214-24. doi: 10.1037/a0036053. Epub 2014 Mar 10. PMID 24611691
- [Result] Manne SL, Siegel S, Kashy D, Heckman CJ. Cancer-specific Relationship Awareness, Relationship Communication, and Intimacy Among Couples Coping with Early Stage Breast Cancer. J Soc Pers Relat. 2014 May;31(3):314-334. doi: 10.1177/0265407513494950. PMID 25242854
- [Result] Manne, S. & Ostroff, J. (2011). Couple-focused group intervention for women diagnosed with early stage breast cancer and their partners. In. D. Kissane & M Watson (Eds.), IPOS Academy Handbook of Psychotherapies in Cancer Care. (pp. 129-139). Chichester, UK: Wiley.